CLINICAL TRIAL: NCT06649747
Title: A Double-blind, Placebo-controlled, Multi-center Phase II Study of the Safety, Tolerability, Efficacy and Pharmacokinetics of Oral AFA-281 in Patients With Painful Lumbosacral Radiculopathy
Brief Title: Safety and Efficacy Study on AFA-281 for the Treatment of Low Back Pain
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Afasci Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFA-281-202
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lumbosacral Radiculopathy
Keywords: Analgesics; Inflammatory pain; Neurologic Diseases; Neuromuscular Diseases; Neuropathic pain,; Peripheral Nervous System Diseases
MeSH Terms: conditions — Nervous System Diseases; Neuromuscular Diseases; Neuralgia; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low dose (Active Comparator): Name: AFA-281; Dosage Form: 5 and 20mg; Dosage: 60mg daily three times a day (TID) for 28 consecutive days
  Interventions: Drug: AFA-281
- Mid Dose (Active Comparator): Name: AFA-281; Dosage Form: 5 and 20mg; Dosage: 120 mg daily three times a day for 28 consecutive days
  Interventions: Drug: AFA-281
- High Dose (Active Comparator): Name: AFA-281; Dosage Form: 5 and 20mg; Dosage: 240 mg daily three times a day for 28 consecutive days
  Interventions: Drug: AFA-281
- Placebo (Placebo Comparator): Name: Placebo Dosage form: matching study drug Dosage: 0 mg daily three times a day for 28 consecutive days
  Interventions: Drug: AFA-281

INTERVENTIONS:
Drug: AFA-281 — A small molecule, orally available

SUMMARY:
The goal of this clinical trial is to evaluate if the drug candidate AFA-281 works to treat chronic low back and leg pain caused by painful lumbosacral radiculopathy (PLSR) in adults. This trial will also evaluate the safety of AFA-281. The main questions it aims to answer are:

* Does AFA-281 mitigate pain?
* What are the side effects (if any)? Researchers will compare AFA-281 to a placebo (a look-alike substance that contains no drug) to see if AFA-281 works to treat chronic low back and leg pain.

Participants will:

* Take drug AFA-281 or a placebo three times every day for 4 weeks
* Visit the clinic once every 2 weeks for checkups and tests
* Keep a diary of their pain scores and about mood and sleep questionnaires, and the number of times they use a rescue pain medicines.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter Phase II study of the efficacy, safety, tolerability, and PK of oral AFA-281 in 300 patients with painful lumbosacral radiculopathy (PLSR). Patients will be randomized in to the placebo group or doses of AFA-281, titrated over 2 weeks to reach planned daily doses for Weeks 3 and 4. Trials will be conducted simultaneously at 3 sites to meet enrollment targets. The primary efficacy endpoint is 24-hour average pain score based on the 0-10-point Numeric Pain Rating Scale (NPRS) and key secondary endpoint is Oswestry Disability Index (ODI), rates of adverse events, and PK, among others.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) indicating that the subject has been informed of the procedures to be followed, the experimental nature of the therapy, potential benefits, side effects, risks, and discomforts
2. Men or nonpregnant, non-breastfeeding women 18 to 65 years of age who can read and understand written and spoken local language
3. Clinical diagnosis of CLBP due to LSR in a dermatomal pattern (L4, L5, or S1) that has been present for at least 3 months at the time of screening.
4. MRI imaging is done within 12 months before screening that does not provide evidence of exclusionary pathology (see exclusion criteria). CT is acceptable for subjects with contra-indications for MRI.
5. Willing to discontinue current pain medications from 2 weeks before randomization until the end of the clinical study (treatment).
6. Numeric rating scale (NRS) ≥4 and ≤9 at screening based on the Patient's Global Impression of Severity (PGI-S)

Exclusion Criteria:

1. Neuropathic pain due to other causes rather than LSR (e.g. painful diabetic neuropathy, other neuropathy, spinal abscess, infection, hematoma or malignancy; phantom limb pain)
2. Has a history of peripheral neuropathy (e.g., due to diabetes, alcohol consumption, other causes, or idiopathic) or evidence of peripheral neuropathy upon neurological examination
3. History of surgical intervention for LSR at the radicular level of the current pain episode.
4. Current indication for neurosurgery (e.g. progressive motor loss due to compression) or planned surgical intervention for LSR within the duration of the study
5. Has planned surgical intervention for PLSR within the duration of the study. (Subjects with persistent radicular pain after prior surgery are eligible.)
6. Spinal stenosis with neurogenic claudication (pain present during walking and signs of significant lumbar stenosis on existing MRI or CT scan)
7. Presence of spinal cord stimulator.
8. Hypersensitivity/allergic reaction to other T-type calcium agents, such as (but not limited to) ethosuximide, zonisamide, and the mixed sodium and T-type calcium channel blocker lamotrigine and .
9. Patients who failed a relatively adequate treatment with a tricyclic antidepressants (TAC), selective serotonin reuptake inhibitors (SSRIs) and serotonin and norepinephrine reuptake inhibitors (SNRIs)
10. Concurrent illnesses that would be a contraindication to trial participation, including, but not limited to:

    1. Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before screening
    2. New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled hypertension
    3. Clinically significant electrocardiographic (ECG) abnormality per the investigator assessment
    4. Has a history or risk of seizures or a history of epilepsy, clinically significant head injury, or related neurological disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2027-04-01 (Estimated); Primary Completion 2032-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 2 weeks baseline and 4 weeks of treatment, and 2 weeks after the end of treatment
  On a scale of 0 to 10, with 0 being no pain at all and 10 being the worst pain imaginable
Safety- Number of Participants with Treatment-Related Adverse Events (AEs) | Baseline (2 weeks) and 4 weeks of the treatment, and 4 weeks of followup
  AEs will be assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Tmax | Predose and Day 28
  Blood samples collected and analyzed for Tmax
Cmax | Predose and Day 28
  Blood samples collected and analyzed for Cmax
Half life | Predose and Day 28
  Blood samples collected and analyzed for half life
AUC | Predose and Day 28
  Blood samples collected and analyzed for AUC

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Xie, MD, PhD, Study Director — Afasci Inc

IPD SHARING:
Plan to Share IPD: No